CLINICAL TRIAL: NCT06650553
Title: Clinical Study on Umbilical Cord Blood-Supported Haploidentical Hematopoietic Stem Cell Transplantation for the Treatment of Aplastic Anemia
Brief Title: Umbilical Cord Blood-Supported Haplo-HSCT for Aplastic Anemia Treatment Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-018-FS02
Record Dates: First submitted 2024-09-28; First posted 2024-10-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2024-09

CONDITIONS: Aplastic Anemias
Keywords: Aplastic Anemias; Stem Cell Transplantation; Umbilical Cord Blood
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Umbilical Cord Blood-Supported Haplo-HSCT for Aplastic Anemia Treatment Study (Experimental): In patients with AA undergoing hematopoietic stem cell transplantation, the feasibility of the umbilical cord blood combined with haploidentical transplantation scheme is assessed by comparing it with sibling fully matched transplantation using a non-inferiority analysis method (with the time of neutrophil engraftment after transplantation as the primary efficacy indicator). At the same time, indicators such as the time of platelet engraftment, infection incidence (including CMV, EBV incidence), acute/chronic GvHD incidence, transplant-related mortality (TRM), event-free survival (EFS), and overall survival (OS) are monitored to evaluate the safety and effectiveness of this scheme.
  Interventions: Procedure: Clinically diagnosed AA patients are divided into HLA-matched HSCT group and umbilical cord blood-supported haplo-HSCT group.

INTERVENTIONS:
Procedure: Clinically diagnosed AA patients are divided into HLA-matched HSCT group and umbilical cord blood-supported haplo-HSCT group. — Conditioning regimen consisted of the following1)Severe aplastic anemia(SAA):FC-ATG:Flu 30 mg/m^2/d ×4d (- 7d- -4d), CTX 22.5 -25mg/kg/d × 4d (-7d- -4d), ATG 7.5mg in total（- 5d- -2d).2)Transfusion-dependent non-severe aplastic anemia（TD-NSAA) and Paroxysmal nocturnal hemoglobinuria (PNH) acquired clonal-aplastic anemia(AA):BU/FC-ATG:Bu 0.8mg/kg(q6h -8d）+FC-ATG. The GVHD prophylaxis program was Application of Anti-CD25 Humanized Monoclonal Antibody 50mg (+1d,+4d);cyclosporine A + mycophenolate mofetil (MMF)+short course methotrexate (MTX).The infusion time of umbilical cord blood (UCB) stem cells in the UCB-assisted haploidentical hematopoietic stem cell transplantation (UCB-Haplo-HSCT) group: 4 hours before the infusion of peripheral blood stem cells.In the follow-up phase, outcome evaluation indicators must be collected according to the follow-up plan, ensuring data quality.

SUMMARY:
Aplastic anemia (AA) is a rare bone marrow failure syndrome with an annual incidence of about 0.74/100,000, affecting all ages but more common in the elderly. It's divided into congenital and acquired forms, with the latter being more prevalent. The primary acquired form is linked to T lymphocyte activation and genetic factors. The best treatment is allogeneic hematopoietic stem cell transplantation (allo-HSCT), with a near 90% cure rate. Sibling allo-HSCT is ideal but finding a match is challenging. For those who relapse after immunosuppressive therapy, haploidentical HSCT is a viable option despite risks like graft failure and GVHD. Advances in transplantation have made haplo-HSCT's efficacy comparable to other methods. Recent studies suggest co-transplantation with umbilical cord blood cells can improve outcomes by hastening hematopoietic recovery and prognosis. Our study will evaluate the feasibility and safety of this approach in AA treatment, comparing it to sibling fully matched transplantation, with a focus on infection rates, GVHD incidence, TRM, and EFS, aiming to enhance treatment practices and benefit patients and the medical industry.

DETAILED DESCRIPTION:
Aplastic anemia (aplastic anaemia，AA) is a syndrome of bone marrow hematopoietic dysfunction （bone marrow hematopoietic failure，BMF）with an annual incidence rate of approximately 0.74/100,000 people, affecting all age groups with a higher incidence rate in the elderly, and similar incidence rates between males and females. AA is divided into congenital and acquired types, with acquired AA being more common. The pathogenesis of primary acquired AA is mainly related to the abnormal activation of T lymphocytes, and genetic background may also play a role in the development and progression of AA. Currently, allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the best treatment for AA, with a cure rate close to 90%. Sibling allogeneic hematopoietic stem cell transplantation (HLA-matched HSCT) is the preferred treatment plan, but it is not easy to find a fully matched sibling donor. For patients who relapse after immunosuppressive therapy (IST), haploidentical hematopoietic stem cell transplantation (haplo-HSCT) is a good alternative, despite the risks of engraftment failure, infection, and graft-versus-host disease (GVHD). With the advancement of transplantation technology, the efficacy of haplo-HSCT is not significantly different from that of unrelated donor hematopoietic stem cell transplantation (MUD-HSCT) and HLA-matched sibling donor hematopoietic stem cell transplantation (MSD-HSCT). Studies have shown that haplo-HSCT has a higher survival rate in treating patients with severe aplastic anemia (SAA), and there is no significant difference compared to MSD-HSCT.To address the risk of complications associated with haplo-HSCT, recent research has indicated that co-transplantation with third-party umbilical cord blood cells can shorten the time for hematopoietic reconstitution and improve prognosis. The co-transplantation of third-party umbilical cord blood with bone marrow and peripheral blood hematopoietic stem cells has become a new transplantation option. Studies at home and abroad have shown that combined third-party transplantation can shorten the time for hematopoietic reconstitution and improve long-term survival rates. This study plans to adopt a prospective, open-label, parallel-controlled trial design to conduct a clinical study of non-related umbilical cord blood-assisted haploidentical allogeneic hematopoietic stem cell transplantation for the treatment of AA. The study will compare the umbilical cord blood combined with haploidentical transplantation plan with sibling fully matched transplantation, to assess the feasibility and safety of the umbilical cord blood combined with haploidentical transplantation plan, and to monitor the incidence of patient infections, acute/chronic GVHD incidence, transplant-related mortality (TRM), and event-free survival (EFS), in the hope of providing new practical experience in the field of AA treatment, and bringing dual benefits to patients and the social medical enterprise.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 6-75 years
* Patients diagnosed with Severe Aplastic Anemia (SAA) , Transfusion-Dependent Non-Severe Aplastic Anemia (TD-NSAA) or Paroxysmal nocturnal hemoglobinuria (PNH) acquired clonal-aplastic anemia(AA) according to the Chinese Guidelines for the Diagnosis and Treatment of Aplastic Anemia (2022 Edition) and suitable for allo-HSCT
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time to neutrophil engraftment | 60 days
  Neutrophil engraftment was defined as the first of three consecutive days on which the patient's absolute neutrophil count was 500/uL.

SECONDARY OUTCOMES:
Time to platelet engraftment | 60 days
  It was defined as independence from platelet transfusion for at least 7 days with a platelet count of more than 20 × 10^9/L.
Incidence of infections (including CMV and EBV incidence) | 100 days,6 months,12 months,24 months
  CMV DNAemia was defined as positive CMV-DNA in the blood when the copies exceeded 500 copies/ml.EBV DNAemia was defined as positive EBV-DNA in the blood when the copies exceeded 500 copies/ml.
Overall survival rate (OS) | 24 months
  Overall survival is a secondary endpoint that will be measured as time from the start of treatment until death from any cause, or the last date the patient was known to be alive.
Event-free survival (EFS) | 24 months
  Considering as event aGVHD, SOS, relapse and death
Incidence of acute/chronic GvHD | 24 months
  aGVHD (acute GVHD) was defined according to the 1994 Consensus Conference on Acute GVHD Grading and graded from I to IV. Chronic GVHD (cGVHD) was graded as limited or extensive.
Transplant-related mortality (TRM) | 100 days,6 months,12 months,24 months
  Transplant-related mortality (TRM) is defined as the proportion of patients who die as a direct or indirect result of the complications arising from the hematopoietic stem cell transplantation (HSCT) process, rather than from the underlying disease for which the transplant was performed. This includes deaths due to graft failure, severe infections, organ toxicity, graft-versus-host disease (GVHD), and other treatment-related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, Dr., Study Director — Shanxi Bethune Hospital Regulatory Authority
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China